CLINICAL TRIAL: NCT06025175
Title: Low Level Lazer Therapy Effect on Vertebral Artery Blood Flow in Elderly With Cervical Disc Degeneration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Shymaa yussuf abo zaid, Lecturer, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T_int_08/2023_519
Record Dates: First submitted 2023-08-20; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Disc Degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: Two groups Group (A) and group(B)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lazer group (Experimental): 30 patients will receive low level lazer therapy 3 times per week for 12 weeks.
  Interventions: Radiation: Low level Lazer therapy; Other: Routine exercises
- Control group (Other): 30 patients will receive only exercises.
  Interventions: Other: Routine exercises

INTERVENTIONS:
Radiation: Low level Lazer therapy — 30 patients will receive low level lazer therapy 3 times a week for 12 weeks.
  Arms: Lazer group
Other: Routine exercises — 30 patients will receive only routine exercises 3 times a week for 12 weeks.

SUMMARY:
This study will include 60 elderly patients with cervical disc degeneration, from both gender who are aged from 60 - 75 years old.

DETAILED DESCRIPTION:
The 60 patients will divided into two groups, with 30 patients in each group. group(A): will receive low level lazer and exercises for three times per week for 12 weeks.

Group (B): will receive only exercises. Resistivity index of both right and left vertebral arteries will be measured before and after the 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. elderly patients with age range between 60 and 75 years old.
2. with cervical disc degeneration.

Exclusion Criteria:

1. patients with uncontrolled hypertension.
2. Patients with uncontrolled diabetes mellitus.
3. Patients with severe cardiac or chest diseases.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Resistivity index of both right and left vertebral arteries | 12 weeks
  Resistivity index of both right and left vertebral arteries will be measured before and after the 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Shymaa yussuf abo zaid, Qina, Egypt